CLINICAL TRIAL: NCT02774746
Title: Gastroschisis Outcomes of Delivery (GOOD) Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Amy Wagner, Professor, Pediatric Surgery, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 898740-1
Record Dates: First submitted 2016-05-11; First posted 2016-05-17 (Estimated); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Gastroschisis
MeSH Terms: conditions — Gastroschisis | interventions — Parturition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 35-week delivery group (Active Comparator): Subjects to be delivered at 35 0/7 weeks through 35 6/7 weeks.
  Interventions: Other: 35-week delivery
- 38-week delivery group (Active Comparator): Subjects to be expectantly managed to spontaneous delivery, delivered by 38 0/7 weeks through 38 6/7 weeks.
  Interventions: Other: 38-week delivery

INTERVENTIONS:
Other: 35-week delivery — Induction at 35 weeks gestational age
  Arms: 35-week delivery group
Other: 38-week delivery — Observation to spontaneous delivery or induction at 38 weeks gestational age
  Arms: 38-week delivery group

SUMMARY:
The objective of this study is to investigate the hypothesis that delivery at 35 0/7- 35 6/7 weeks in stable patients with gastroschisis is superior to observation and expectant management with a goal of delivery at 38 0/7 - 38 6/7 weeks. To test this hypothesis, we will complete a randomized, prospective, multi-institutional trial across NAFTNet-affiliated institutions. Patients may be enrolled in the study any time prior to 33 weeks, but will be randomized at 33 weeks to delivery at 35 weeks or observation with a goal of 38 weeks. The primary composite outcome will include stillbirth, neonatal death prior to discharge, respiratory morbidity, and need for parenteral nutrition at 30 days.

DETAILED DESCRIPTION:
Gastroschisis is the most common congenital abdominal wall abnormality in which the intestines are outside of body floating in the amniotic fluid. This is diagnosed by prenatal ultrasound at 18-20 weeks gestation. Gastroschisis occurs in 1 out of every 4000 births and the incidence is increasing. The majority of patients with gastroschisis have an uncomplicated neonatal course and recover well after surgical repair. However, subsets of gastroschisis patients have more complicated courses due to loss of intestine or blockages of the intestine These infants have a higher risk of death and long-term morbidity. Additionally, gastroschisis patients have an increased risk of in-utero fetal demise or stillbirth.

The potential risk of pregnancy loss late in the third trimester has prompted some physicians to deliver gastroschisis patients prior to term. This results in an increased chance of additional prematurity-related complications. There is no consensus about the ideal time to deliver a baby with gastroschisis and practice patterns vary widely. It is unclear which offers the fetus a chance at a better outcome: early delivery to mitigate risk of stillbirth and intestinal injury versus delivery closer to term.

Retrospective data published show inconsistent results on outcomes with early delivery or later gestational age delivery in gastroschisis. There have been two randomized, prospective trials with delivery early versus awaiting spontaneous labor. The first included 42 patients rendering the study largely underpowered. There was a trend towards decreased length of hospital stay and earlier time to full enteral feeding in the early delivery group, but this did not reach statistical significance. The latest study was stopped early because of futility and an increased risk of sepsis in the early group. There was no increase in sepsis in the early group in the first trial, and the study design of this trial varies greatly from both studies.

Standard delivery times for uncomplicated gastroschisis are between 34 and 39 weeks gestation. As the current available literature does not adequately answer the question of optimal gestational age of delivery in patients with gastroschisis, the objective of this study is to investigate the hypothesis that delivery at 35 0/7 - 35 6/7 weeks in stable patients with gastroschisis is superior to observation and expectant management with a goal of delivery at 38 0/7 - 38 6/7 weeks. To test this hypothesis, we will complete a randomized, prospective, multi-institutional trial. Patients may be enrolled in the study any time prior to 33 weeks but will be randomized at 33 weeks to delivery at 35 weeks or observation with a goal of 38 weeks. The primary outcome will be based on a weighted composite comprised of intrauterine fetal demise, neonatal/infant death prior to discharge, respiratory morbidity, gastrointestinal morbidity, and sepsis. We will compare the rates of the composite outcome as well as the individual components to determine whether a significant difference between the two strategies can be detected. Secondary maternal outcomes include need for labor induction, need for cesarean section, and complications of delivery including infection, blood transfusions, and thromboembolic events. We will also evaluate antenatal test values, such as amniotic fluid index, estimated fetal weight, and intra- and extra-abdominal bowel dilation. Secondary neonatal outcomes include birth and discharge weight, central venous catheter days, sepsis, intestinal atresia, necrotizing enterocolitis, time to enteral autonomy, individual components of respiratory morbidity, need for caffeine, and length of stay.

Given the unprecedented patient data being collected for the randomized trial, we plan to leverage the infrastructure built for this study to generate the largest prospective, multicenter database of gastroschisis-related (maternal, fetal, and neonatal) outcomes in the United States. The database will provide data for future development of both hypotheses and study design regarding gastroschisis-related outcomes. The associated biobank will collect blood from the neonatal participants to be stored and analyzed in future research.

ELIGIBILITY:
Inclusion criteria:

To be eligible for study inclusion, subjects are required to meet the following criteria:

1. Speak English or Spanish
2. Age of ≥18 years old
3. Have a diagnosis of an isolated fetal gastroschisis confirmed via sonogram at ≤33 weeks gestation
4. Have a singleton pregnancy
5. Capable of providing written informed consent for study participation
6. Established Estimated Date of Confinement (EDC) prior to 22 0/7 weeks GA by last menstrual period (LMP) with ultrasound confirmation or ultrasound dating when LMP is unknown.

Exclusion criteria:

Subjects will be excluded from enrollment for any of the following criteria

1. Fetal anomaly unrelated to gastroschisis, such as a chromosomal abnormality or another congenital structural abnormality (if known; no additional testing required for research participation)
2. Severe intrauterine growth restriction / fetal growth restriction (defined as growth below the 5th percentile for gestational age)
3. Maternal history of previous stillbirth (intrauterine fetal demise)
4. Maternal history of spontaneous preterm (<36 weeks) delivery
5. Maternal cervical length < 25 mm prior to 24 weeks of gestation if documented
6. Maternal hypertension
7. Maternal insulin-dependent diabetes
8. Prenatal care initiated after 24 weeks of gestation
9. An active case of COVID-19 (confirmed by a positive test for COVID-19) that is not recovered (confirmed by a negative test for COVID-19) by the date of randomization
10. Unstable pregnancy defined as meeting any of the following criteria

    1. Abnormal amniotic fluid volume defined as oligohydramnios or polyhydramnios where the maximal vertical pocket (MVP) is < 2 cm or > 8 cm in the third trimester, respectively
    2. Umbilical artery Dopplers with S/D ratio or resistive index (RI) > 97th percentile for age with or without absent or reversed end diastolic flow
    3. Non-stress test (NST) or biophysical profile (BPP) deemed non-reassuring by treating clinician
11. Concurrent enrollment in another study that requires either a treatment or intervention which would either alter the delivery plan or potentially influence the maternal, fetal, and neonatal outcomes of this study
12. Traditional surrogacy, gestational surrogacy, gestational carrier, or gestational surrogate
13. Incapable of providing informed consent
14. Are not their own legally authorized representative.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2018-02-23 (Actual); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of the proportion of the primary composite outcome (occurrence of any of the 3 clinical risks: IUFD, neonatal death, and sepsis) between groups as estimated from the ITT population. | Date of consent until NICU Discharge. Discharge dates for patients vary and depend on each individual's recovery progress, medical needs, and overall condition. In general, this entire time frame can take up to 30 weeks.
  The primary outcome is the composite endpoint combining the following three clinical risks: (1) intrauterine fetal demise, (2) neonatal/infant death prior to neonatal intensive care unit (NICU) discharge, (3) sepsis.
  The probability of the composite endpoint will be compared between groups as defined by the ITT population using a one-sided test at a 2.3% nominal significance level for the alternative hypothesis that the experimental early delivery group has lower probability of the composite endpoint compared to term delivery group. The nominal significance level will be adjusted based on the timing of the interim analysis if different from the original plan. The Wald test for two proportions will be used. We will report the estimated difference in the probabilities along with the Wald confidence interval using the nominal significance level.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Wagner, MD, Principal Investigator — Medical College of Wisconsin
Locations (38):
- United States (38):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Loma Linda University Children's Hospital, Loma Linda, California
  - Lucile Packard Children's Hospital Stanford, Stanford, California
  - Children's Hospital of Colorado, Aurora, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Nemours Children's Hospital, Delaware, Wilmington, Delaware
  - University of South Florida & Tampa General Hospital, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Riley Children's Hospital, Indianapolis, Indiana
  - Norton Healthcare, Inc., Lousiville, Kentucky
  - University of Maryland, Baltimore, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Brigham and Women's Hospital & Boston Children's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - CS Mott Children's & Von Voigtlander Women's Hospital, Michigan Medicine, Ann Arbor, Michigan
  - Children's MN, Midwest Fetal Care Center, Minneapolis, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - St. Louis University, SSM Health Cardinal Glennon Children's Hospital & SSM Health St. Mary's Hospital, St Louis, Missouri
  - Washington University in St. Louis & St. Louis Children's Hospital, St Louis, Missouri
  - Columbia University Irving Medical Center, New York, New York
  - New York Presbyterian - Weill Cornell Medicine, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - University of North Carolina Hospitals, Chapel Hill, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Women & Infants Hospital/Rhode Island Hospital (Hasbro Children's), Providence, Rhode Island
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Cook Children's Medical Center, Fort Worth, Texas
  - University of Texas Medical Branch Galveston, Galveston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - The Woman's Hospital of Texas / Obstetrix Maternal-Fetal Medicine Specialists of Houston, Houston, Texas
  - Christus Children's / Baylor College of Medicine, San Antonio, Texas
  - University of Utah & Primary Children's Hospital, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - University of Wisconsin - Madison, Madison, Wisconsin
  - Medical College of Wisconsin & Children's Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided
Plan to share data if NIH funded.